CLINICAL TRIAL: NCT02910024
Title: Theta-Burst-Stimulation in Der frühen Rehabilitation Von Schlaganfallpatienten
Brief Title: Theta-Burst-Stimulation in Early Rehabilitation of Stroke
Acronym: TheSiReS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Gereon R. Fink, Prof. Dr. med., University of Cologne
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Uni-Koeln-1778; U1111-1172-6026 (Other: WHO); CIV-15-09-013868 (Other: EUDAMED); DRKS00008963 (Registry Identifier: DRKS)
Record Dates: First submitted 2016-09-08; First posted 2016-09-21 (Estimated); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Clinical Protocols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real-rTMS (Active Comparator): Repetitive transcranial magnetic stimulation (rTMS) of the primary motor cortex in the lesioned hemisphere using the intermittent theta-burst-stimulation protocol (iTBS; application of 3 pulses with a frequency of 50 Hz, in a theta-rhythm of 5 Hz for 2 seconds, repeated every 10 seconds, duration of one session: about 3,5 minutes) before physiotherapy for 8 days
  Interventions: Device: Magstim Super Rapid2 System, intermittent theta-burst-stimulation (iTBS) protocol
- Sham-rTMS (Sham Comparator): Repetitive transcranial magnetic stimulation (rTMS) in sham position (tilted coil over parieto-occipital vertex) before physiotherapy for 8 days
  Interventions: Device: Magstim Super Rapid2 System, sham-stimulation (in iTBS)

INTERVENTIONS:
Device: Magstim Super Rapid2 System, intermittent theta-burst-stimulation (iTBS) protocol — iTBS applied over ipsilesional M1
  Arms: Real-rTMS
Device: Magstim Super Rapid2 System, sham-stimulation (in iTBS) — iTBS applied with tilted coil over parieto-occipital vertex
  Arms: Sham-rTMS

SUMMARY:
The present prospective, randomized, controlled, double-blinded trial investigates the effects of intermittent theta-burst stimulation (iTBS) during the early rehabilitation after stroke. Patients with hemipresis will receive either sham or real iTBS over their affected hemispheres before occupational therapy for 8 days. Motor recovery is assessed one day after the intervention phase and three months after enrollment.

DETAILED DESCRIPTION:
To date, rehabilitation of stroke with hemiparesis mainly includes physiotherapy and occupational therapy. Yet, the majority of patients retain movement impairment relevant for activities of daily living. One explanation for this deficit is the insufficient recovery of connectivity between brain regions after stroke. It is possible to modulate this process by repetitive transcranial magnetic stimulation (rTMS) using the protocol of intermittent theta-burst stimulation (iTBS). Previous data indicate that modulation of the motor cortex with iTBS enhances the effects of subsequent motor training. The present study aims at investigating whether daily repetitive transcranial magnetic stimulation over 8 days combined with subsequent physiotherapy leads to better motor recovery, compared with physiotherapy after sham stimulation. In the first weeks and after three months, motor function, degree of disability and quality of life are examined in order to evaluate the effects of iTBS in the rehabilitation of stroke patients.

Amendment (approved by the Ethics-Committee of the Medical Faculty of the University of Cologne, 20/12/2016): Specification of exclusion criteria.

Amendment (approved by the Ethics-Committee of the Medical Faculty of the University of Cologne, 15/11/2018): Change of inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* written consent
* age: 40-90 years
* ischemic stroke
* hemiparesis with impaired hand motor function

Exclusion Criteria:

* Subjects who are legally detained in an official institute (§20 MPG)
* Participation in clinical trial within the last 12 weeks
* Electronic implants or ferromagnetic Implants located in the head, neck or thorax (e.g. clips, intracranial shunt, artificial heart valve, pacemaker)
* Medication pump (e.g. insulin pump)
* Metal splinters in eye or head
* Pregnancy / breastfeeding
* Severe Neurodegenerative disease
* Severe Neuroinflammatory disease
* History of seizures / epilepsy
* Physical addiction to alcohol, medication, or drugs (excluded: nicotine)
* Insufficient compliance
* Present or past malignant tumor involving the central nervous system
* Severe Psychiatric disease
* Clinically manifest bilateral hemiparesis or infarcts in the primary motor cortex or along the tractus corticospinalis in the hemisphere ipsilateral to the hemiparesis
* Pre-existing cerebral infarctions with hemiparesis or pre-existing cerebral infarctions in the primary motor cortex or along the tractus corticospinalis, excluding microangiopathic changes (e.g. clinically asymptomatic lacunae <1cm)
* Known brain lesion (surgical, traumatic)
* Evidence for enhanced cerebral pressure
* Severe cardial dysfunction
* life expectancy < 12 months
* NIHSS Score > 20
* Blood glucose imbalances resistant to treatment (<50 mg/dl or >300 mg/dl)
* Elevated blood pressure resistant to treatment (RR > 185/110mmHg)
* Systemic Thrombolysis using r-tPA or thrombectomy within the last 24 hours before enrollment in study
* Medication with benzodiazepines, high-potency antipsychotics or tricyclic antidepressants before hospitalization or long-term during hospitalization

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Relative grip force | 3 months after enrollment
  grip force as measured with vigorimeter

SECONDARY OUTCOMES:
Relative grip force | after 8 days of intervention, and 3 months after enrollment
  grip force as measured with vigorimeter
Motor function | after 8 days of intervention, and 3 months after enrollment
  Action Research Arm Test, ARAT
Motor function | after 8 days of intervention, and 3 months after enrollment
  Fugl-Meyer Motor Scale of the upper extremity, FM
Stroke severity | after 8 days of intervention, and 3 months after enrollment
  National Instituts of Health Stroke Scale, NIHSS
Degree of disability | after 8 days of intervention, and 3 months after enrollment
  modified Rankin Scale, mRS
Motorcortex excitability | after 8 days of intervention, and 3 months after enrollment
  Motor evoked potential induced by stimulation of the affected motor cortex, MEP
Motorcortex excitability | after 8 days of intervention, and 3 months after enrollment
  Resting motor threshold as measured by stimulation of the affected motor cortex, RMT
Quality of life | after 8 days of intervention, and 3 months after enrollment
  EuroQol 5D questionnaire, EQ-5D
Activities of daily living at admission and discharge in external rehabilitation facility | 3 months after enrollment
  Barthel-Index (BI) scores as documented by external rehabilitation facility
Days of rehabilitation after intervention phase | 3 months after enrollment
  Days of rehabilitation after intervention phase as documented by external rehabilitation facility

CONTACTS AND LOCATIONS:
Overall Officials: Gereon R Fink, Univ.-Prof. Dr., Principal Investigator — University of Cologne
Locations (1):
- Klinik und Poliklinik für Neurologie, Universitätsklinikum Köln, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hensel L, Grefkes C, Tscherpel C, Ringmaier C, Kraus D, Hamacher S, Volz LJ, Fink GR. Intermittent theta burst stimulation applied during early rehabilitation after stroke: study protocol for a randomised controlled trial. BMJ Open. 2019 Dec 30;9(12):e034088. doi: 10.1136/bmjopen-2019-034088. PMID 31892668